CLINICAL TRIAL: NCT03867097
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Phase 2 Pilot Study Evaluating Intravenous Iloprost in Subjects With Symptomatic Raynaud's Phenomenon Secondary to Systemic Sclerosis
Brief Title: Intravenous Iloprost in Subjects With Symptomatic Raynaud's Phenomenon Secondary to Systemic Sclerosis (Phase 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Civi Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES-201
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Raynaud Phenomenon Secondary to Systemic Sclerosis
Keywords: systemic sclerosis; raynaud phenomenon
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line. Study drug will be initiated at a starting dose 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Interventions: Drug: Placebo IV infusion
- Iloprost Injection, for intravenous use (Active Comparator): Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line. Study drug will be initiated at a starting dose 0.5 ng/kg/min up to 2.0 ng/kg/min.
  Interventions: Drug: Iloprost Injection, for intravenous use

INTERVENTIONS:
Drug: Placebo IV infusion — Study drug will be initiated at a starting dose of 0.5 ng/kg/min up to 2.0 ng/kg/min. Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line.
  Arms: Placebo
Drug: Iloprost Injection, for intravenous use — Study drug will be initiated at a starting dose of 0.5 ng/kg/min up to 2.0 ng/kg/min. Subjects will receive study drug for 5 consecutive days as an IV infusion over 6 hours each day via a peripheral line.
  Arms: Iloprost Injection, for intravenous use

SUMMARY:
This is a Phase 2, multicenter, double-blind, randomized, placebo-controlled study to evaluate the effect of iloprost on the symptomatic relief of Raynaud's Phenomenon attacks in subjects with symptomatic Raynaud's Phenomenon secondary to Systemic Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects must be greater than or equal to 18 years of age
* Subjects must have a diagnosis of Systemic Sclerosis
* Subjects must have a diagnosis or history of Raynaud's Phenomenon
* Subjects must have a minimum of 10 symptomatic Raynaud's Phenomenon attacks
* Female subjects of childbearing potential and male subjects must agree to use contraception for the duration of the study
* Subjects must be willing and able to comply with the study requirements and give informed consent for participation in the study

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding
* Subjects with systolic blood pressure <85 mmHg
* Subjects with an estimated glomerular filtration rate <30 mL/min/1.73 m2
* Subjects with Child-Pugh Class B or Class C liver disease or an alanine aminotransferase and/or aspartate aminotransferase value >3 × the upper limit of normal at screening.
* Subjects with gangrene, digital ulcer infection, or requirement of cervical or digital sympathectomy
* Subjects with intractable diarrhea or vomiting
* Subjects with a risk of clinically significant bleeding events including those with coagulation or platelet disorders
* Subjects with a history of major trauma or hemorrhage
* Subjects with clinically significant chronic intermittent bleeding such as active gastric antral vascular ectasia or active peptic ulcer disease
* Subjects who have had any cerebrovascular events
* Subjects with a history of myocardial infarction or unstable angina within 6 months of screening
* Subjects with acute or chronic congestive heart failure
* Subjects with a history of life-threatening cardiac arrhythmias
* Subjects with a history of hemodynamically significant aortic or mitral valve disease
* Subjects with more than mild restrictive or congestive cardiomyopathy uncontrolled by medication or implanted device.
* Subjects with known pulmonary hypertension, pulmonary arterial hypertension, or pulmonary veno-occlusive disease
* Subjects with a history of significant restrictive lung disease defined as forced vital capacity <45% predicted and diffusing capacity of the lungs for carbon monoxide <40% predicted (uncorrected for hemoglobin).
* Subjects with a history of cervical or digital sympathectomy
* Subjects with scleroderma renal crisis
* Subjects with a concomitant life-threatening disease with a life expectancy <12 months
* Subjects who have a clinically significant disorder, that in the opinion of the Investigator, could contraindicate the administration of study drug, affect compliance, interfere with study evaluations, or confound the interpretation of study results
* Subjects who have taken or are currently taking any parenteral, inhaled, or oral prostacyclin or prostacyclin receptor agonists
* Subjects must not initiate dosing of oral, topical, or intravenous (IV) vasodilators or if currently receiving any vasodilator must have been stably medicated
* Subjects with any history of acetaminophen intolerability
* Subjects with any malignancy that requires treatment during the study period, that has required treatment within 1 year of screening, or that is currently not in remission.
* Subjects who have used any investigational medication or device for any indication within 30 days or 5 half-lives (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Benton, Pharm D, Study Director — Civibio Pharma, Inc.
Locations (16):
- United States (16):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Pacific Arthritis Care Center of Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Georgetown University Medical Center - Department of Rheumatology, Washington D.C., District of Columbia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Toledo Medical Center (UTMC) - Ruppert Health Center, Toledo, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Houston - Division of Rheumatology and Clinical Immunogenetics, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Arthritis Northwest Rheumatology PLLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated on 07 March 2019 and completed on 06 August 2019. It was conducted in 16 sites located in the United States.
Pre-assignment Details: In this study 41 participants with Systemic Sclerosis (SSc) were screened.34 participants who had at least 10 symptomatic Raynaud's phenomenon (RP) attacks on the 5-day eligibility period were randomized on to the study: 17 to the placebo arm and 17 to the Iloprost arm.
Period: Overall Study
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.59) | 50.2 (13.48) | 49.6 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 13 | 16 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Phosphodiesterase inhibitor at baseline [Number; unit: n (%)]
  Yes | 7 | 5 | 12
  No | 10 | 12 | 22
Weekly frequency of symptomatic RP attacks at baseline [Median (Standard Deviation); unit: no. of attacks] | 42.32 (29.635) | 37.05 (18.643) | 39.69 (24.525)

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Symptomatic RP Attacks
Description: The primary efficacy parameter is the change in the weekly frequency of symptomatic RP attacks from baseline.
  The baseline weekly frequency of symptomatic RP attacks was defined as the average number of weekly symptomatic RP attacks that occurred during the 10- to 25-day baseline ePRO diary completion period.
  The double-blind endpoint weekly frequency of symptomatic RP attacks was defined as the average number of weekly symptomatic RP attacks that occurred during Days 8 to 21, inclusive.
Time Frame: Day 8 - Day 21 will be compared to baseline
Population: The modified Intention-to-Treat (mITT) Population was defined as all randomized subjects who initiated infusion of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of RP attacks per week
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
Number analyzed (Participants) | 17 | 17
Number of RP attacks per week | -14.32 [-20.15 to -8.48] | -15.09 [-21.14 to -9.04]
Statistical Analysis 1: Comparison: Placebo vs Iloprost Injection, for Intravenous Use; Treatment comparison of change versus placebo. LS mean difference in change. When a subject had no RP attacks in the past 24 hours, the frequency was considered as zero for that day. The LS means, SEs, CIs, and p-values came from an ANCOVA model with randomized treatment group and use of phosphodiesterase inhibitors at screening (yes, no) as factors and baseline as a covariate; Test type: Superiority; p = 0.8498, ANCOVA; LS mean difference in change = -0.77, 95% CI 2-sided [-9.04 to 7.49], Standard Error of Mean 4.047 — The Shapiro-Wilk normality test of residuals indicated that the data did not have a normal distribution (p-value 0.0108)
Statistical Analysis 2: Comparison: Placebo vs Iloprost Injection, for Intravenous Use; Change in the Weekly Frequency of Symptomatic Raynaud's Phenomenon Attacks From Baseline to the Double-Blind Endpoint Using Nonparametric Analysis - Modified Intent-to-Treat Population. Treatment comparison of change versus placebo; Test type: Superiority; p = 0.9729, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.24, 95% CI 2-sided [-9.97 to 9.32]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 35
Arm/Group | Placebo | Iloprost Injection, for Intravenous Use
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 14/17 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Iloprost Injection, for Intravenous Use (N=17)
Headache (Nervous system disorders) | 5 (5) | 16 (16)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Infusion site pain (General disorders) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Vessel puncture site pruritus (General disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 5 (5)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03867097/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03867097/SAP_001.pdf